CLINICAL TRIAL: NCT06530134
Title: Promote Awareness of the Driving Abilities of Post-stroke Patients: Interest of On-board Cameras and Self-assessment Questionnaires During a Driving Situation.
Brief Title: Promote Awareness of the Driving Abilities of Post-stroke Patients.
Acronym: AUTOCAM-AVC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Mutualiste de Rééducation et de Réadaptation Fonctionnelles de Kerpape (Other)
Collaborators: University Gustave Eiffel (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2020-A03377-32
Record Dates: First submitted 2021-10-20; First posted 2024-07-31 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Cerebrovascular Accident
Keywords: post-stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: This research is part of a Research Involving the Human Person of the interventional with minimal risks and constraints type (RIPH2).This is a prospective, monocentric, comparative, randomized and controlled study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- With video feedback (Experimental): Activation of on-board cameras during driving situation.
  Interventions: Other: Driving situation and video feedback
- Without video feedback (Other): Non-Activation of on-board cameras during driving situation.
  Interventions: Other: Driving situation and usual recommendations (without video feedback)

INTERVENTIONS:
Other: Driving situation and video feedback — At the end of the driving situation, 35 patients will be asked to express themselves and analyze 4 driving situations resulting from the course of the driving situation using video feedback.
  Arms: With video feedback
Other: Driving situation and usual recommendations (without video feedback) — At the end of the driving situation, 35 patients will be asked to express themselves and analyze 4 driving situations resulting from the course of the driving situation without video feedback, according to the usual recommendations.
  Comparison of responses to all questionnaires and interview grids sent before and after driving, to patients and professionals will determine whether video feedback promotes awareness of the difficulties of driving post-stroke patients.
  Arms: Without video feedback

SUMMARY:
Patients with cerebrovascular accident (CVA) may present with a deficit of awareness of the disorders which results in a lack of correct self-estimation of their own abilities and difficulties in terms of both cognition and driving. It is therefore important to develop tools to help professionals take this deficit into account in their driving assessments and also to help patients better identify their real abilities.

This research project thus proposes a protocol making it possible to promote decision-making whether or not to resume driving by multidisciplinary teams.

The main objective is to determine to what extent video feedback promotes awareness of the ability to manage post-stroke patients, compared to a group of control patients receiving the usual recommendations.

ELIGIBILITY:
Inclusion Criteria:

* Stroke (ischemic and / or hemorrhagic) between 1 month and 6 months
* Holder of a driving license for more than 3 years
* No resumption of driving
* MoCA score ≥ 10
* Affiliation to a social security scheme or beneficiary of such a scheme
* Having signed a free, informed and written consent
* Medically stable

Exclusion Criteria:

* Aphasia with severe comprehension disturbances, severe hemineglect, unstable epilepsy, severe visual disturbances (binocular vision <6/10, visual field <120 ° in binocular, <50 ° to the right and to the left beyond the central point, <30 ° vertically.
* History of neurological disease responsible for cognitive impairment
* Need for vehicle modifications except automatic gearbox
* Subject being in a period of exclusion from another protocol
* Insufficient command of the French language
* Protected adults (curators)
* Pregnancy declared
* Being unable to issue their consent

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2021-10-12 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Awareness of driving behavior. | Day 0
  This criterion will be measured using the difference between patient's and the professional's scores from the interview with the situation analyzes.
  If the difference between the patient's score and that of the professionals is close to zero, it means that the patient correctly self-estimates their driving abilities. If the difference is positive, it means the patient overestimates their abilities. If the difference is negative, it means the patient underestimates their abilities.
  The professionals score is the mean of the score of each professional (occupational therapist and driving instructor)
  The patient fills out the questionnaire before and after the interview. The two professionals fill out the questionnaire once, before the interview. This score of driving behavior awareness after the interview will be compared to that before the interview, reflecting any potiential change in awareness following the interview.

SECONDARY OUTCOMES:
The concordance between the opinion of the two professionals (driving instructor and occupational therapist) and that of the patient about returning to driving, then compare this concordance between the two arms. | Day 0
  The score of question 4 of the "Q final-pro" questionnaire will be compared to question 7 of the "Q final-pa" questionnaire (with or without feedback depending on the arm). The differences between the two opinions (Patient Opinions-Professional Opinions) on all the evaluations will allow to establish a score "of concordance of the opinions of rework". A score equal to zero means that the opinions are the same between the patient and the professionals (best outcome), a positive or negative score means that the opinions are divergent. The closer the score is to zero, the better the result. The same process will be followed with the control group that did not receive video feedback in order to compare the concordance scores of the rework notices between the two arms.
The concordance between the opinion of the driving teacher and the occupational therapist after the on-road test | Day 0
  Study of the concordance between the total score of the TRIP (Test Ride for Investigating Practical Fitness to Drive) grid (Qpost-cond-trip) of the driving teacher and that of the occupational therapist (score/100)
  Calcul of a correlation coefficient : the higher the coefficient, the more consistent the assessments between the 2 professionals are (better outcome).
The concordance between the opinion of the driving teacher and the occupational therapist for the interview grid | Day 0
  Study of the concordance between the total score of the interview grid (Qentr-pro) of the driving teacher and that of the occupational therapist (score/28).
  Calcul of a correlation coefficient : the higher the coefficient, the more consistent the assessments between the 2 professionals are (better outcome).
Compare the MOCA score between patients who had a favorable opinion (PFO) and patients who had an unfavorable opinion (PUO) | Day 0
  • [MOCA test /30 score] PFO compared to PUO (MOCA : Montreal Cognitive Assessment)
Compare the score of Rey's Figure between patients who had a favorable opinion (PFO) and patients who had an unfavorable opinion (PUO) | Day 0
  • [Rey's Figure score /36, execution time (s)] PFO compared to PUO
Compare the score of Bell Test between patients who had a favorable opinion (PFO) and patients who had an unfavorable opinion (PUO) | Day 0
  • [Bell Test score /35, execution time (s)] PFO compared to PUO
Compare the attentional performance between patients who had a favorable opinion (PFO) and patients who had an unfavorable opinion (PUO) | Day 0
  TAP Scores PFO compared to PUO (TAP : Attention Assessment Tests)
Compare the information processing speed between patients who had a favorable opinion (PFO) and patients who had an unfavorable opinion (PUO) | Day 0
  • Score combining the scores at the code and symbol tests /38 ] PFO compared to PUO (WAIS : Wechsler Adult Intelligence Scale)
Compare the working memory performance between patients who had a favorable opinion (PFO) and patients who had an unfavorable opinion (PUO) | Day 0
  • [WAIS-IV digit memory score /19] PFO compared to PUO
Links between cognitive performance and the awareness score of driving skills. | Day 0
  To study the links between cognitive performance and awareness, MOCA score will be correlated with awareness scores (Patient Score Difference - Professional Score obtained before the interview (Qentr-pro completed before the interview)).
Links between awareness of cognitive impairment and awareness of driving skills. | Day 0
  To assess awareness of cognitive disorders, the difference in scores (Patient Score / Self-assessment - Professional Score / Hetero-assessment) of the BRIEF A will be calculated.
  The Brief A test (Behavior Rating Inventory of Executive Function) aims to investigate the existence of a deficit of consciousness of cognitive disorders in patients. The patient's assessment score from the self-assessment questionnaire will be compared with that of professionals (hetero-assessment). The difference between the two scores (Patient Score / Self-assessment - Average Professional Score / Hetero-assessment) will determine whether the patient has a lack of awareness of his cognitive disorders. If the difference (Patient Score - Professional Score) is positive, the patient overestimates his disorders; if it is negative, the patient underestimates them; if it is zero it means that the patient is estimating them correctly.
Become patients at 6 months | At 6 months
  The behaviors and driving strategies of patients 6 months after their resumption of driving (Q follow-up) will be compared with those declared in the initial questionnaire on the answers to the following questions: "Since you have resumed driving, do you think that you have more difficulty driving than before? "," If so, in which situations do you think you have more difficulty "," Since your recovery, do you think you are avoiding more situations than before? "," If so, what are the situations you think you can avoid the most? "," Since your recovery, have you developed different driving strategies for driving? "," If so, what strategies have you put in place to drive safely "," Since your recovery, has the activity of driving scared you more than before? "," Do you think the activity of driving is more tiring than before? "
Acceptability of the video device by professionals and patients | Day 0
  The acceptability of the video device by professionals will be measured by the answers obtained to question 6 of the final questionnaire completed by professionals (Qfinal-pro) (e.g. questions: as a professional, having video feedback was easy to use during the interview, choice of items to tick). The closer the score is to 12, the higher the acceptability of the video device by professionals.
  The acceptability of the video device by the patients will be measured thanks to the feelings that the patients will have expressed in question 2 of the final questionnaire (on interest, pleasure, stress, perceived usefulness, satisfaction and pleasure experienced by compared to the device).

CONTACTS AND LOCATIONS:
Overall Officials: Pauline Coignard, Doctor, Principal Investigator — CMRRF de Kerpape
Locations (1):
- CMRRF de Kerpape, Ploemeur, Brittany Region, France

IPD SHARING:
Plan to Share IPD: No